CLINICAL TRIAL: NCT04945733
Title: A Phase 2, Open-label Study of Amivantamab in Subjects With Previously Treated Advanced or Metastatic Gastric or Esophageal Cancer
Brief Title: A Study of Amivantamab in Participants With Previously Treated Advanced or Metastatic Gastric or Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to reconsideration of development strategy
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109026; 61186372GIC2001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amivantamab: Gastric Cancer (GC) Cohorts (Experimental): Participants in Phase 2a GC cohorts will receive intravenous (IV) infusion of weight-based dose of amivantamab in 28-day cycles. Participants with body weight less than (<) 80 kilograms (kg) will receive IV infusion of amivantamab 1,050 milligrams (mg) and participants with body weight greater than or equal to (>=) 80 kg will receive IV infusion of amivantamab 1,400 mg once weekly in Cycle 1 and then every 2 weeks in subsequent cycles (on Days 1 and 15 of each cycle), followed by additional dosing based on body weight if recommended by clinical trial management team (CTMT) (amivantamab 1750 mg for body weight <80 kg and 2100 mg for body weight >=80 kg as IV infusion) every 2 weeks on Days 1 and 15 of 28 day cycle. Phase 2b GC expansion cohorts will be initiated if activity is observed within Phase 2a cohorts.
  Interventions: Drug: Amivantamab
- Amivantamab: Esophageal Cancer (EC) Cohorts (Experimental): Participants in Phase 2a EC cohorts will receive IV infusion of weight-based dose of amivantamab in 28-day cycles. Participants with body weight <80 kg will receive IV infusion of amivantamab 1,050 mg and participants with body weight >=80 kg will receive IV infusion of amivantamab 1,400 mg once weekly in Cycle 1 and then every 2 weeks in subsequent cycles (on Days 1 and 15 of each cycle) followed by additional dosing based on body weight if recommended by CTMT (amivantamab 1750 mg for body weight <80 kg and 2100 mg for body weight >=80 kg as IV infusion) every 2 weeks on Days 1 and 15 of 28 day cycle. Phase 2b EC expansion cohorts will be initiated if activity is observed within Phase 2a cohorts.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered intravenously.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this study is to investigate the activity of amivantamab in gastric cancer (GC) and esophageal cancer (EC) participants (Phase 2a), and to characterize the preliminary antitumor activity of amivantamab in selected GC and EC population (Phase 2b).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed gastric (including gastroesophageal junction [GEJ]) or esophageal cancer (EC) that is locally advanced, unresectable, or metastatic, and not eligible for curative treatment
* Participant must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. If only 1 measurable lesion exists, it may be used for the screening biopsy if the baseline tumor assessment scans are performed greater than or equal to (>=) 7 days after the biopsy
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Gastric or GEJ Cancer Only - Must be refractory or ineligible to at least 2 prior lines of standard of care systemic therapy. Prior therapies must include fluoropyrimidine- and platinum-based chemotherapy. Participants with known human epidermal growth factor receptor (HER) 2 expression must have had HER2 targeting therapy as part of the prior therapy

Esophageal Cancer Only

- Must be refractory or intolerant to at least 1 prior line of systemic therapy. Prior therapies must include fluoropyrimidine-, and platinum-based chemotherapy (including chemoradiation therapy given as stage intravenous [IV] setting)

Exclusion Criteria:

* Participant has an uncontrolled illness, including but not limited to the following: diabetes; ongoing or active bacterial infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week before enrollment]), symptomatic viral infection, or any other clinically significant infection; active bleeding diathesis and psychiatric illness/social situation that would limit compliance with study requirements
* Participant has received prior epidermal growth factor receptor (EGFR) or tyrosine-protein kinase mesenchymal-epithelial transition (cMet)-directed therapies
* Participant has had prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks or 4 half-lives whichever is longer or had radiation therapy within 4 weeks before the first administration of study treatment. For agents with long half-lives, the maximum required time since last dose is 28 days. Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less, (except for alopecia or post-radiation skin changes [any grade], Grade less than or equal to [<=] 2 peripheral neuropathy, and Grade <=2 hypothyroidism stable on hormone replacement)
* Participant has untreated brain metastases (a participant with definitively, locally treated metastases who is clinically stable, asymptomatic, and off corticosteroid treatment for at least 2 weeks prior to the first administration of study treatment is eligible), history of leptomeningeal disease or spinal cord compression that has not been treated definitively with surgery or radiation. If brain metastases are diagnosed on screening imaging, the participant may be rescreened for eligibility after definitive treatment
* Participant has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening. Esophageal cancer participants with history of completely resolved radiation pneumonitis (defined as radiographically stable for 3 months prior to enrollment without need of any treatment) may be enrolled

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (10):
- Japan (10):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - Saitama Cancer center, Kitaadachi-gun
  - Niigata Cancer Center Hospital, Niigata
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Osaka University Hospital, Suita-shi
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Yokohama City University Medical Center, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 cohorts: Phase 2a cohorts (including Phase 2a extension cohort) and Phase 2b expansion cohort in participants with previously treated advanced or metastatic gastric or esophageal cancer. However, due to study termination, no participants were enrolled in Phase 2a extension cohorts and Phase 2b cohorts. Hence the results were only presented for Phase 2a cohorts.
Groups:
- Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg): Participants with previously treated advanced or metastatic gastric/gastroesophageal junction cancer (GC) exhibiting varying degrees of epidermal growth factor receptor (EGFR), tyrosine-protein kinase mesenchymal-epithelial transition (MET), or both as determined by immunohistochemistry (IHC) received amivantamab 1050 milligrams (mg) for body weight less than (<) 80 kilograms (kg) or 1400 mg for body weight greater than or equal to (>=) 80 kg as an intravenous (IV) infusion in each 28-day cycles. During Cycle 1, amivantamab was administered once weekly on Days 1, 8, 15 and 22 with first dose split over Day 1 (350 mg) and Day 2 (700 mg for body weight <80 kg/1050 mg for body weight >=80 kg). From Cycle 2 onwards, amivantamab was administered on Days 1 and 15 until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death whichever comes first. Participants were followed up for safety up to 30 days after the last dose.
- Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg): Participants with previously treated advanced or metastatic esophageal cancer (EC) exhibiting varying degrees of EGFR, MET, or both as determined by IHC received amivantamab 1050 mg for body weight <80 kg or 1400 mg for body weight >=80 kg as an IV infusion in each 28-day cycles. During Cycle 1, amivantamab was administered once weekly on Days 1, 8, 15 and 22 with the first dose split over Day 1 (350 mg) and Day 2 (700 mg for body weight <80 kg or 1050 mg for body weight >=80 kg). From Cycle 2 onwards, amivantamab was administered on Days 1 and 15 until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death whichever comes first. Participants were followed up for safety up to 30 days after the last dose.
- Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg): Participants with previously treated advanced or metastatic EC exhibiting varying degrees of EGFR, MET, or both as determined by IHC received amivantamab 1750 mg for body weight <80 kg or 2100 mg for body weight >=80 kg as an IV infusion in each 28-day cycles. During Cycle 1, amivantamab was administered once weekly on Days 1, 8, 15 and 22 with the first dose split over Day 1 (350 mg) and Day 2 (1400 mg for body weight <80 kg or 1750 mg for body weight >=80 kg). From Cycle 2 onwards, amivantamab was administered on Days 1 and 15 until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death whichever comes first. Participants were followed up for safety up to 30 days after the last dose.
Period: Overall Study
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Started | 29 | 30 | 3
Completed | 25 | 24 | 3
Not Completed | 4 | 6 | 0
Not completed — Physician Decision | 1 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Total
Number analyzed (Participants) | 29 | 30 | 3 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 18 | 2 | 33
  >=65 years | 16 | 12 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.97) | 62.7 (10.35) | 60 (9) | 63.2 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 0 | 11
  Male | 24 | 24 | 3 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 30 | 3 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 29 | 30 | 3 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 29 | 30 | 3 | 62

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: ORR was defined as the percentage of participants who achieved a confirmed complete response (CR) or partial response (PR) as determined by investigator per RECIST version 1.1. As per RECIST version 1.1, CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<)10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-progressive disease (PD). For non-target lesions, PD: unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression.
Time Frame: From start of the treatment (Day 1) up to 30 days after the last dose of study drug (up to 9 months)
Population: Response evaluable analysis set included all participants who received at least 1 dose of study treatment, met all eligibility criteria for the study and had a baseline and at least 1 post-baseline efficacy disease assessments, or had disease progression/death due to disease progression prior to the first post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 23 | 28 | 2
Percentage of Participants | 4.3 [0.1 to 21.9] | 10.7 [2.3 to 28.2] | 0 [0.0 to 84.2]

2. Secondary Outcome: Disease Control Rate (DCR) Per RECIST Version 1.1
Description: DCR was defined as the percentage of participants achieving CR or PR or stable disease (SD) for at least 6 weeks as defined by RECIST version 1.1. As per RECIST version 1.1 CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR was defined as >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. For non-target lesions, PD: unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, and no appearance of new lesion(s).
Time Frame: From start of the treatment (Day 1) up to 30 days after the last dose of study drug (up to 9 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 23 | 28 | 2
Percentage of Participants | 26.1 [10.2 to 48.4] | 67.9 [47.6 to 84.1] | 100 [15.8 to 100]

3. Secondary Outcome: Duration of Response (DOR) as Per RECIST Version 1.1
Description: DOR was defined as time between date of first documented response (CR/PR) and date of first documented progression or death, whichever occurred first. CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes short axis measures <10 mm. PR was defined as >=30% decrease in sum of measures (tumor lesions-longest diameter and nodes-short axis) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. For non-target lesions, PD: unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. There was no participant who had event (CR/PR) in Phase 2a EC higher dose cohort, hence data could not be collected and analyzed for this cohort.
Time Frame: From the date of first documented response up to date of first documented PD or death (up to 9 months)
Population: Response evaluable analysis set included all participants who received at least 1 dose of study treatment, met all eligibility criteria for study and had a baseline and at least 1 post-baseline efficacy disease assessments, or had disease progression/death due to disease progression prior to first post-baseline disease assessment. Here 'N' (overall number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 1 | 3 | 0
Months | NA [NA to NA] — Here, 'NA' signifies that median, lower and upper limit of 95% confidence interval (CI) could not be calculated due to less number of participants with events. | 2.86 [2.79 to NA] — Here, 'NA' signifies that upper limit of 95% CI could not be calculated due to less number of participants with events. |

4. Secondary Outcome: Time to Response (TTR) as Per RECIST Version 1.1
Description: TTR was defined as time from date of first amivantamab administration to date of achieving objective response (CR/PR) as assessed by investigator per RECIST v1.1 among participants who achieved objective response. Per RECIST v1.1, CR: disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. For non-target lesions, PD: unequivocal progression of existing non-target lesions. The appearance of one or more new lesions was also considered progression. There was no participant who had event (CR/PR) in Phase 2a EC higher dose cohort, hence data could not be collected and analyzed for this cohort.
Time Frame: From first dose of study treatment until first documentation of CR or PR (up to 9 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 1 | 3 | 0
Months | 1.45 [NA to NA] — Here, 'NA' signifies that lower and upper limit of 95% CI could not be calculated due to less number of participants with events. | 1.41 [1.41 to NA] — Here, 'NA' signifies that upper limit of 95% CI could not be calculated due to less number of participants with events. |

5. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from the date of first dose of study drug until the date of objective disease progression or death (by any cause in the absence of progression), whichever comes first, based on investigator assessment using RECIST Version 1.1.
Time Frame: From day of first dose (Day 1) until PD or death (up to 9 months)
Population: All treated analysis set included all participants who took at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 29 | 30 | 3
Months | 1.45 [1.41 to 1.48] | 4.11 [2.10 to 4.17] | 2.99 [1.41 to NA] — Here, 'NA' signifies that upper limit of 95% CI could not be calculated due to less number of participants with events.

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs was defined as AEs occurring at or after first dose of study drug up to 30 days after last dose or until the start of new anticancer therapy, whichever occurred first. TEAEs were graded according to NCI-CTCAE v5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE. All TEAEs including serious and non-serious events are reported in this outcome measure.
Time Frame: From start of the treatment (Day 1) up to 30 days after last dose or start of new anticancer therapy, whichever occurred first (up to 9 months)
Population: The safety analysis set included all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 29 | 30 | 3
Participants
  Grade 1 | 4 | 3 | 1
  Grade 2 | 14 | 17 | 1
  Grade 3 | 8 | 9 | 1
  Grade 4 | 0 | 0 | 0
  Grade 5 | 3 | 1 | 0

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Amivantamab
Description: Cmax was defined as the maximum observed serum concentration of amivantamab. The concentrations of amivantamab were measured using a validated, specific, and sensitive enzyme-linked immunosorbent assay (ELISA) method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for Cmax was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 24, 26, 48, 72, 96 and 168 hours post-dose on Day 1 of Cycle 1; pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: The pharmacokinetics (PK) analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement. Here 'N' (overall number of participants analyzed) = participants evaluable for this outcome measure and 'n' (number analyzed) = refers to participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (mcg/mL)
Groups:
- Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg): Participants with previously treated advanced or metastatic GC and EC exhibiting varying degrees of EGFR, MET, or both as determined by IHC received amivantamab 1050 mg for body weight <80 kg or 1400 mg for body weight >=80 kg as an IV infusion in each 28-day cycles. During Cycle 1, amivantamab was administered once weekly on Days 1, 8, 15 and 22 with the first dose split over Day 1 (350 mg) and Day 2 (700 mg for body weight <80 kg or 1050 mg for body weight >=80 kg). From Cycle 2 onwards, amivantamab was administered on Days 1 and 15 until disease progression, unacceptable toxicity, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death whichever comes first. Participants were followed up for safety up to 30 days after the last dose.
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 13 | 12 | 0 | 25
Micrograms per milliliter (mcg/mL)
  Cycle 1 Day 1 | 356 (91.6) | 370 (78.2) |  | 363 (84.0)
  Cycle 2 Day 1: number analyzed (Participants) | 8 | 10 | 0 | 18
  Cycle 2 Day 1 | 820 (221) | 866 (196) |  | 845 (202)

8. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for Amivantamab
Description: Tmax was defined as the time to reach maximum observed serum concentration of amivantamab. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for Tmax was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: as for outcome 7
Population: The PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement. Here 'N' (overall number of participants analyzed) = participants evaluable for this outcome measure and 'n' (number analyzed) = refers to participants evaluable at specified time points.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 13 | 12 | 0 | 25
Hours (h)
  Cycle 1 Day 1 | 28.42 [27.02 to 31.00] | 29.65 [28.80 to 31.62] |  | 29.23 [27.02 to 31.62]
  Cycle 2 Day 1: number analyzed (Participants) | 8 | 10 | 0 | 18
  Cycle 2 Day 1 | 4.23 [2.42 to 24.63] | 2.53 [2.27 to 4.53] |  | 3.46 [2.27 to 24.63]

9. Secondary Outcome: Area Under the Curve From Time (0) to Time (168h) (AUC [0-168h]) for Amivantamab
Description: AUC (0-168h) was defined as area under the serum concentration time-curve from time zero to the time point 168 hours. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for AUC (0-168h) was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 24, 26, 48, 72, 96 and 168 hours post-dose on Day 1 of Cycle 1 (each cycle was of 28 days)
Population: The PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement. Here 'N' (overall number of participants analyzed) refers to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms*hours/milliliter (mcg*hr/mL)
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 12 | 12 | 0 | 24
micrograms*hours/milliliter (mcg*hr/mL) | 30990 (8346) | 31548 (7854) |  | 31269 (7930)

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Amivantamab
Description: Area under the serum concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 336 hours was reported. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for AUCtau was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micrograms*hours/milliliter (mcg*hr/mL)
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 4 | 8 | 0 | 12
micrograms*hours/milliliter (mcg*hr/mL) | 137806 (19006) | 162171 (45328) |  | 154049 (39369)

11. Secondary Outcome: Phase 2a Gastric Cancer and Esophageal Cancer Cohorts: Serum Trough Concentrations (Ctrough) of Amivantamab
Description: Ctrough of amivantamab in GC and EC cohorts were reported. Ctrough was defined as pre-dose serum drug concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]).
Time Frame: Pre-dose at 0 hour: Days 8 and 15 of Cycle 1; Days 1 and 15 of Cycles 2, 3 and 4; Day 1 of Cycles 6 and 8 (each cycle was of 28 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 24 | 28 | 52
Micrograms per milliliter (mcg/mL)
  Pre-dose Cycle 1 Day 8: number analyzed (Participants) | 12 | 12 | 24
  Pre-dose Cycle 1 Day 8 | 119 (34.9) | 136 (45.1) | 128 (40.5)
  Pre-dose Cycle 1 Day 15 | 214 (73.7) | 222 (74.6) | 218 (73.5)
  Pre-dose Cycle 2 Day 1: number analyzed (Participants) | 21 | 27 | 48
  Pre-dose Cycle 2 Day 1 | 308 (99.5) | 342 (77.4) | 327 (88.5)
  Pre-dose Cycle 2 Day 15: number analyzed (Participants) | 10 | 21 | 31
  Pre-dose Cycle 2 Day 15 | 231 (85.6) | 259 (80.7) | 250 (82.0)
  Pre-dose Cycle 3 Day 1: number analyzed (Participants) | 5 | 16 | 21
  Pre-dose Cycle 3 Day 1 | 166 (86.6) | 234 (58.5) | 217 (70.3)
  Pre-dose Cycle 3 Day 15: number analyzed (Participants) | 4 | 15 | 19
  Pre-dose Cycle 3 Day 15 | 154 (83.3) | 210 (87.1) | 198 (87.1)
  Pre-dose Cycle 4 Day 1: number analyzed (Participants) | 3 | 12 | 15
  Pre-dose Cycle 4 Day 1 | 105 (73.2) | 236 (82.8) | 210 (95.4)
  Pre-dose Cycle 4 Day 15: number analyzed (Participants) | 1 | 11 | 12
  Pre-dose Cycle 4 Day 15 | 139.0 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant. | 203 (54.1) | 198 (54.8)
  Pre-dose Cycle 6 Day 1: number analyzed (Participants) | 1 | 3 | 4
  Pre-dose Cycle 6 Day 1 | 122.3 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant. | 190 (35.7) | 173 (44.7)
  Pre-dose Cycle 8 Day 1: number analyzed (Participants) | 1 | 1 | 2
  Pre-dose Cycle 8 Day 1 | 111.4 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant. | 100.0 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant. | NA (NA) — Here, 'NA' signifies that, per planned analysis, data was not summarized where number of participants analyzed was less than 3. Only individual participant data was collected and analyzed which is reported in the first 2 arms.

12. Secondary Outcome: Phase 2a Esophageal Cancer Higher Dose Cohort: Serum Trough Concentrations (Ctrough) of Amivantamab
Description: Ctrough of amivantamab in phase 2a EC higher dose cohort was reported. Ctrough was defined as pre-dose serum drug concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose at 0 hour: Day 15 of Cycle 1; Days 1 and 15 of Cycles 2 and 3; Day 1 of Cycles 6 and 8 (each cycle was of 28 days)
Population: The PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement. Here 'N' (overall number of participants analyzed) = the participants evaluable for this outcome measure and 'n' (number analyzed) = participants evaluable at specified time points. As planned participant wise data was collected and analyzed when "n" was less than (<) 3.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 2
Micrograms per milliliter (mcg/mL)
  Pre-dose Cycle 1 Day 15: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 1 Day 15: Participant 1 | 333 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 1 Day 15: Participant 2: number analyzed (Participants) | 1
  Pre-dose Cycle 1 Day 15: Participant 2 | 337 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 2 Day 1: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 2 Day 1: Participant 1 | 657 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 2 Day 1: Participant 2: number analyzed (Participants) | 1
  Pre-dose Cycle 2 Day 1: Participant 2 | 779 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 2 Day 15: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 2 Day 15: Participant 1 | 590 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 2 Day 15: Participant 2: number analyzed (Participants) | 1
  Pre-dose Cycle 2 Day 15: Participant 2 | 604 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 3 Day 1: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 3 Day 1: Participant 1 | 433 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 3 Day 1: Participant 2: number analyzed (Participants) | 1
  Pre-dose Cycle 3 Day 1: Participant 2 | 600 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 3 Day 15: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 3 Day 15: Participant 1 | 460 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 6 Day 1: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 6 Day 1: Participant 1 | 295 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Pre-dose Cycle 8 Day 1: Participant 1: number analyzed (Participants) | 1
  Pre-dose Cycle 8 Day 1: Participant 1 | 314 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.

13. Secondary Outcome: Phase 2a Gastric Cancer Cohort: Terminal Elimination Half-Life (t1/2) for Amivantamab
Description: Terminal elimination half-life (t1/2) was the time measured for the serum concentration of a drug to decrease by half of its initial concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method.
Time Frame: Pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: The PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement. Here 'N' (overall number of participants analyzed) = the participants evaluable for this outcome measure and 'n' (number analyzed) = participants evaluable at specified row. As planned participant wise data was collected and analyzed when "n" was <3.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 2
Hours
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 226.0 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 264.5 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant.

14. Secondary Outcome: Phase 2a Esophageal Cancer and Overall Combined Cohorts: Terminal Elimination Half-Life (t1/2) for Amivantamab
Description: Terminal elimination half-life (t1/2) was the time measured for the serum concentration of a drug to decrease by half of its initial concentration. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for EC cohort and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for t1/2 was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 7 | 0 | 9
Hours | 254.7 (43.0) |  | 252.6 (38.7)

15. Secondary Outcome: Apparent Clearance at Steady State (CLss) of Amivantamab
Description: Clearance was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for CLss was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liters/hour (L/h)
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 4 | 8 | 0 | 12
Liters/hour (L/h) | 0.00775 (0.00122) | 0.00695 (0.00200) |  | 0.00722 (0.00176)

16. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Amivantamab
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for Vss was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: Pre-dose, 0, 2, 24, 48, 72, 168 and 336 hours post-dose on Day 1 of Cycle 2 (each cycle was of 28 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 1 | 6 | 0 | 7
Liters | 3.59 (NA) — Here, 'NA' signifies that standard deviation could not be calculated due to single evaluable participant. | 2.61 (1.04) |  | 2.75 (1.02)

17. Secondary Outcome: Accumulation Ratio (AR) of AUCtau for Amivantamab
Description: Accumulation ratio for AUC was calculated as AUC (0-336h) for Cycle 2 Day 1 divided by AUC (0-168h) for Cycle 1 Day 1. The concentrations of amivantamab were measured using a validated, specific, and sensitive ELISA method. Data for this outcome measure was planned to be collected and analyzed for each cancer type (GC and EC) and overall participants (GC and EC combined cohorts: Amivantamab [1050/1400 mg]). As planned, data for AR of AUCtau was not collected and analyzed for Phase 2a EC higher dose cohort.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) | Overall: Phase 2a GC and EC Combined Cohorts: Amivantamab (1050/1400 mg)
Number analyzed (Participants) | 4 | 8 | 0 | 12
Ratio | 4.32 (0.51) | 5.12 (0.72) |  | 4.85 (0.74)

18. Secondary Outcome: Number of Participants With Anti-Amivantamab Antibodies
Description: Number of participants with anti-amivantamab antibodies were reported. Serum samples were assessed for anti-drug antibodies.
Time Frame: From start of the treatment (Day 1) up to 30 days after the last dose of study drug (up to 9 months)
Population: The immunogenicity analysis set included all participants who received at least 1 dose of study treatment and had at least 1 evaluable post-baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
Number analyzed (Participants) | 26 | 30 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening up to 30 days after last dose of study drug (up to 10 months); Serious AEs and Other AEs: From start of the treatment (Day 1) up to 30 days after last dose of study drug (up to 9 months)
Description: The safety analysis set included all participants who took at least 1 dose of study treatment.
Arm/Group | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg)
All-Cause Mortality (participants affected / at risk) | 5/29 | 2/30 | 0/3
Serious Adverse Events (participants affected / at risk) | 9/29 | 7/30 | 0/3
Other Adverse Events (participants affected / at risk) | 28/29 | 30/30 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) (N=29) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) (N=30) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) (N=3)
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Disease Progression (General disorders) | 2 | 0 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 1 | 0
Retroperitoneal Abscess (Infections and infestations) | 1 | 0 | 0
Kidney Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2a Gastric Cancer Cohort: Amivantamab (1050/1400 mg) (N=29) | Phase 2a Esophageal Cancer Cohort: Amivantamab (1050/1400 mg) (N=30) | Phase 2a Esophageal Cancer Higher Dose Cohort: Amivantamab (1750/2100 mg) (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 1
Stomatitis (Gastrointestinal disorders) | 7 | 4 | 0
Fatigue (General disorders) | 1 | 3 | 0
Malaise (General disorders) | 5 | 5 | 1
Oedema Peripheral (General disorders) | 7 | 5 | 1
Pyrexia (General disorders) | 1 | 3 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2 | 0
Liver Disorder (Hepatobiliary disorders) | 3 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 4 | 3
Paronychia (Infections and infestations) | 5 | 10 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 12 | 13 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 1 | 0 | 1
Weight Decreased (Investigations) | 1 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 6 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 10 | 17 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 9 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Embolism (Vascular disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was planned to be conducted in 2 cohorts: Phase 2a cohorts (including Phase 2a extension cohort) and Phase 2b expansion cohort. However, due to study termination, no participants were enrolled in Phase 2a extension and Phase 2b cohorts. Hence results were only presented for Phase 2a cohorts. Phase 2b specific outcome measure (overall survival) were not included in the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04945733/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT04945733/SAP_001.pdf